CLINICAL TRIAL: NCT06965530
Title: The Role of Medically Tailored Groceries in Mitigating Food Insecurity and Improving Pregnancy Outcomes Through Clinic-Community Partnerships
Brief Title: Nourishing Tomorrow: Role of Medically Tailored Groceries in Addressing Food Insecurity During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University Hospitals Cleveland Medical Center (Other); MetroHealth Medical Center (Other); Greater Cleveland Food Bank (Unknown)
Responsible Party: Principal Investigator, Elaine Borawski, Vice Chair for Applied Research, Department of Nutrition, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY20241029; R01NR021490 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-05-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Prematurity; Birth Outcome, Adverse
Keywords: Randomized trial; Behavioral intervention
MeSH Terms: conditions — Premature Birth; Pregnancy Complications | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinic-Based Medically Tailored Groceries (CB-MTG) (Active Comparator): Standard of Care: Patients enrolled in the health systems clinic-based Food is Medicine Program.
  Interventions: Dietary Supplement: Clinic-Based Medically Tailored Groceries (CB-MTG)
- Home Delivered Medically Tailored Groceries (HD-MTG) (Experimental): Patient received home delivered medically tailored groceries every two weeks during pregnancy and up to 6 months post-delivery.
  Interventions: Dietary Supplement: Home Delivered Medically Tailored Groceries (HD-MTG)
- Home Delivered Medically Tailored Groceries PLUS (HD-MTGPLUS) (Experimental): Same as Arm 2, receiving home delivered medically tailored groceries every two weeks during pregnancy and up to 6 months post-delivery, but receives additional nutrition and culinary education and support throughout the trial.
  Interventions: Dietary Supplement: Home Delivered Medically Tailored Groceries plus Education (HD-MTG_PLUS)

INTERVENTIONS:
Dietary Supplement: Clinic-Based Medically Tailored Groceries (CB-MTG) — Patients have the opportunity to pick up medically tailored groceries every other week at the Food Is Medicine Clinic or Market associated with their provider.
  Arms: Clinic-Based Medically Tailored Groceries (CB-MTG)
Dietary Supplement: Home Delivered Medically Tailored Groceries (HD-MTG) — Patient receive home delivered medically tailored groceries every two weeks during pregnancy and up to 6 months post-delivery.
  Arms: Home Delivered Medically Tailored Groceries (HD-MTG)
Dietary Supplement: Home Delivered Medically Tailored Groceries plus Education (HD-MTG_PLUS) — Patients receive home delivered medically tailored groceries every two weeks during pregnancy and up to 6 months post-delivery, plus also receives additional nutrition and culinary education and support throughout the trial.
  Arms: Home Delivered Medically Tailored Groceries PLUS (HD-MTGPLUS)

SUMMARY:
Medically tailored groceries (MTG), involving grocery items to be prepared at home, selected by a nutritional professional based on a treatment plan, is a growing approach adopted by healthcare systems to address food insecurity in their patient populations, a leading contribution to health disparities such as poor birth outcomes within pregnant populations. However, transportation and other social needs can often hinder patient uptake of clinic-based approaches. Findings from this study will help to better understand how home delivery of MTGs, with and without supplemental education and support to improve food literacy, behavioral and health outcomes.

DETAILED DESCRIPTION:
Medically tailored groceries (MTG) generally involve fresh and shelf-stable grocery items to be prepared at home, selected by a nutritional professional based on a treatment plan and are typically picked up at a clinic, market, or pantry. This clinic-based market or pantry model (CB-MTG) is a growing approach adopted by health care systems in their effort to address food insecurity in their patient population, including University Hospitals of Cleveland (UH) and MetroHealth Medical Center (Metro), two of the three largest health systems in Cleveland, Ohio. Often offered to patients with food-related chronic conditions, CB-MTGs have shown to improve medication adherence, increase fruits and vegetable consumption and decrease HbA1c in people with diabetes. However, less evidence is available on the impact of CB-MTGs with food insecure pregnant individuals, where food insecurity has been strongly associated with prematurity and other negative birth outcomes.

While promising, the CB-MTG approach requires transportation, having the tools and equipment to prepare meals at home and some basic food preparation skills, all potential barriers for low-income pregnant individuals, especially younger parents-to-be or those already with children. The Greater Cleveland Food Bank and partners, seeking to address these barriers, recently developed a home delivered version of MTG (HD-MTG), offered to Medicaid-eligible pregnant individuals across the county, with promising results. The investigators seek to integrate these approaches into patient care for food insecure, pregnant women and test the effectiveness of these two approaches, alongside an additional intervention arm that adds supplemental nutrition and culinary education and support to the home-delivered approach (HD-MTG PLUS). These three approaches will be offered (via randomization) to 360 pregnant individuals (120 per arm) with food insecurity who are patients within UH and Metro's largest urban obstetric practices, each with direct electronic health record (EHR) referral systems to their "food as medicine" clinics/markets. Data are collected at baseline, near/at delivery and 6 months post-delivery. This study seeks to understand the unique contribution of each approach, as well as implementation and intervention uptake barriers, with the goal of building the evidence base of MTG interventions and making recommendations to providers and health systems seeking to address food insecurity and nutrient deficiencies during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Pregnant patients >10 weeks and <22 weeks gestation at randomization (must be consented by 20 weeks)
* Eligible for Medicaid
* Singleton pregnancy, confirmed by ultrasound
* An established patient of the UH or Metro pregnancy clinic
* English speaking
* Lives in Cuyahoga County, Ohio

Exclusion Criteria:

* Under 18 years old

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Food Insecurity | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  6 item, United States Department of Agriculture (USDA) measure; dichotomous outcome
Food Insecurity | Change from baseline to 6-months post delivery
  6 item, USDA measure; dichotomous outcome
Baby Gestational Age | At birth
  Measured in weeks and classified as preterm (<37 weeks) vs. term (37+ weeks)
Baby Birthweight | At birth
  Measured in grams and classified as normal (> or = 2500g), low birth weight (<2500g), very low birthweight (<1500g), extremely low birth weight (<1000g)
Days Hospitalized (Baby) | From date of birth until the date of discharge from the hospital, assessed up to 100 months
  Number of days baby was hospitalized following birth
Neonatal Intensive Care Unit (NICU)/Special Care Nursery (SCN) Utilization | From admission date to the NICU/SCN until the date of discharge from NICU/SCN, assessed up to 100 months
  Number of days baby was admitted to NICU or SCN

SECONDARY OUTCOMES:
Birth Complications | Perioperative/periprocedural
  List of poor maternal and fetal health conditions or outcomes at time of delivery
Prenatal Health Care | From first documented prenatal visit until the baby's delivery date, assessed up to 9 months
  Number / Frequency of prenatal health care visits, extracted from medical record (chart review)
Pregnancy Complications | Perioperative/periprocedural
  Yes / No for any of the following: (1) gestational diabetes; (2)preeclampsia; (3) poor weight gain or loss during pregnancy
Gestational Diabetes Mellitus (GDM) | Assessed up to 40 weeks of pregnancy
  Diagnosis of GDM during pregnancy
Attitudes toward Cooking and Food Preparation | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Mean of 6 items, range 1-5, higher scores indicate more positive attitudes toward cooking
Attitudes toward Cooking and Food Preparation | Change from baseline to 6-months post delivery
  Mean of 6 items, range 1-5, higher scores indicate more positive attitudes toward cooking
Cooking Efficacy | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Mean of 4 items, range 1-5 (not all at confident to extremely confident); higher number indicates higher efficacy; e.g. I can cook nutritious meal; I can cook a meal in a short amount of time; I can cook a nutritious meal without spending a lot of money; I can follow a recipe).
Cooking Efficacy | Change from baseline to 6-months post delivery
  Mean of 4 items, range 1-5 (not all at confident to extremely confident); higher number indicates higher efficacy; e.g. I can cook nutritious meal; I can cook a meal in a short amount of time; I can cook a nutritious meal without spending a lot of money; I can follow a recipe).
Cooking Frequency | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  3 items; from National Health and Nutrition Examination Survey (NHNES); # of times a week cooking breakfast, lunch and dinner
Cooking Frequency | Change from baseline to 6-months post delivery
  3 items; from NHNES; # of times a week cooking breakfast, lunch and dinner
Dietary Quality | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Derived from diet recalls collected with the Nutrition Data System for Research. Includes: total calories, energy density, macronutrient intake, micronutrients, dietary fiber, sugar sweetened beverages, food group intake, and fast food intake
Dietary Quality | Change from baseline to 6-months post delivery
  Derived from diet recalls collected with the Nutrition Data System for Research. Includes: total calories, energy density, macronutrient intake, micronutrients, dietary fiber, sugar sweetened beverages, food group intake, and fast food intake
Healthy Eating Index (HEI) | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Total Healthy Eating Index score, ranging from 1-100, with higher scores indicating higher nutritional quality of diet
Healthy Eating Index (HEI) | Change from Baseline to 6 months post-delivery
  Total Healthy Eating Index score, ranging from 1-100, with higher scores indicating higher nutritional quality of diet
Healthy Eating Self Efficacy (HESE) | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Subscale of the Healthy Eating and Weight Self-Efficacy Scale: Mean of 6 items, range 1-5, higher scores indicate higher level of confidence to choose, prepare and consume healthy food options
Healthy Eating Self-Efficacy (HESE) | Change from Baseline to 6 months post-delivery
  Subscale of the Healthy Eating and Weight Self-Efficacy Scale: Mean of 6 items, range 1-5, higher scores indicate higher level of confidence to choose, prepare and consume healthy food options
Depressive Symptoms | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Edinburgh Perinatal / Postnatal Depression Scale (EDPS); a 10-question survey with each answer given a score of 0-3; higher scores suggest minor or major depression may be present
Depressive Symptoms | Change from baseline to 6-months post delivery
  Edinburgh Perinatal / Postnatal Depression Scale (EDPS); a 10-question survey with each answer given a score of 0-3; higher scores suggest minor or major depression may be present
Perceived Stress | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Mother's stress index score (10-item standardized index, with each answer given a score of 1-5 and higher scores indicating stress is present)
Perceived Stress | Change from baseline to 6-months post delivery
  Mother's stress index score (10-item standardized index, with each answer given a score of 1-5 and higher scores indicating stress is present)
Decision Fatigue | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Decisional Fatigue Scale (DFS) (range 0 to 30; higher total scores are posited to correlate with the intensity of perceived decisional fatigue)
Decision Fatigue | Change from baseline to 6-months post delivery
  Decisional Fatigue Scale (DFS) (range 0 to 30; higher total scores are posited to correlate with the intensity of perceived decisional fatigue)
Social Support | Change from baseline to delivery (assessed up to 40 weeks of pregnancy)
  Multidimensional Scale of Perceived Social Support; 6-item questionnaire, each answer scored 1-5 with higher scores indicating strong social support
Social Support | Change from Baseline to 6 months post-delivery
  Multidimensional Scale of Perceived Social Support; 6-item questionnaire, each answer scored 1-5 with higher scores indicating strong social support

CONTACTS AND LOCATIONS:
Overall Officials: Elaine A Borawski, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals Rainbow Ahuja Women and Children's Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
As required by our National Institute of Nursing Research grant award, please see the required Data Management and Sharing Plan (uploaded as separate document). In brief, at the of the study, de-identified questionnaire, clinical and implementation data will be deposited into the Inter-university Consortium for Political and Social Research (ICPSR) and designated as controlled access. Case Western Reserve University (CWRU) is a member of ICPSR which permits the deposit of data at no charge.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of the primary outcomes paper being published.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT06965530/ICF_000.pdf